CLINICAL TRIAL: NCT00082355
Title: The Treatment of Deep Vein Thrombosis (DVT) of the Lower Extremities With "Low-Dose" Alteplase: a Pilot Study
Brief Title: Low-Dose Alteplase to Treat Blood Clots in Deep Leg Veins
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Richard Chang, M.D. (NIH)
Collaborators: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor-Investigator, Richard Chang, M.D., Senior Clinician, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 040178; 04-CC-0178 (Other: NIH Clinical Center)
Record Dates: First submitted 2004-05-06; First posted 2004-05-06 (Estimated); Results first posted 2012-12-19 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-10

CONDITIONS: Acute Deep Venous Thrombosis of the Lower Extremity
Keywords: r-tPA; Thrombolysis; Clot; Anticoagulation; Fibrinolysis; Deep Vein Thrombosis; DVT
MeSH Terms: conditions — Venous Thrombosis | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alteplase (r-tPA) (Experimental): Patients with DVT of lower extremity will receive up to 4 treatments low dose (<10 mg/day) intraclot injections of alteplase. Intention is to evaluate safety and efficacy of this treatment, and durability of outcomes (for 6 months)in 25 patients.
  Interventions: Drug: Alteplase (Activase, Genentech)

INTERVENTIONS:
Drug: Alteplase (Activase, Genentech) — Dose of Alteplase will not exceed 10 mg/d/leg and is delivered in a concentration of 100ug/mL. The actual dose delivered is based upon the length of the thrombosed vein and 1 mL is injected directly into each centimeter of a thrombosed vein in a lower extremity. The treatment will be repeated up to 4 times over a 4 day period.

SUMMARY:
This study will test the effectiveness of low-dose recombinant tissue plasminogen activator (rtPA, or alteplase) in dissolving blood clots in deep leg veins. Alteplase is used to clear blood clots in coronary arteries in patients having heart attacks. Blood clots can develop in the deep leg veins causing pain and swelling and may break loose and lodge in the lungs. Current routine treatments use anticoagulants such as heparin stop the clots from enlarging and prevent clots from moving to the lung but do not reliably dissolve clots in the leg.In an earlier study we showed that rtPA could be used to actually dissolve the clots. This study will determine whether lower doses of rtPA can dissolve clots with fewer bleeding complications than the current higher-dose regimens.

Patients 18 years of age and older who have blood clots in a deep vein of the pelvis or leg may be eligible for this study if they have had symptoms for 14 days or less and if they have never had clots in their deep veins before.

Participants are admitted to hospital for up to 5 days. On the first treatment day, the patient has a venogram to show the location of the clots. The radiologist injects an x-ray contrast material into a small vein in the foot and watches the dye by x-ray as it moves up the leg, revealing the clot(s). A catheter (plastic tube) is then inserted into a vein either behind the knee, in the groin, or in the neck, and advanced until it reaches the clots. When the catheter is in place, rtPA is injected while the radiologist watches the vein under the x-ray image. The amount of rtPa needed will depends on the size of the clot. Up to five venograms may be done if the clot requires the maximum four rtPA treatments allowed in this study. During the treatments, patients receive standard doses of heparin, given continuously by vein, After completion of treatments, anticoagulation is continued through use of a low molecular weight heparin (usually enoxaparin) given by subcutaneous injection as a transition medication during conversion to anticoagulation with warfarin ( also known as coumadin), another blood thinner, taken by mouth. Patients continue taking warfarin for 6 months.

During thrombolytic therapy, blood samples are drawn shortly before the first dose of rtPA and at five time points afterward to measure the rtPA in the circulation and other factors that indicate whether the rtPA is affecting clotting ability. Blood also is drawn at least once a day to monitor heparin levels.

To evaluate the impact of treatment on the function of the leg, patients return to the Rehabilitation Medicine Department and Radiology department at about 6 weeks (4 to 8 week ) and 6 months for clinical and imaging evaluation of impact of therapy on venous function.

The objectives are to determine how well this treatment will restore venous function and whether this can be done safely- without causing bleeding complications, which have been the main risks of previous thrombolytic treatments.

DETAILED DESCRIPTION:
Deep venous thrombosis (DVT) of the lower extremities is routinely treated with anticoagulants, which is very effective in preventing pulmonary embolism, but does not reliably restore venous function in the leg affected by DVT,often leaving permanent vein damage that leads to chronic disability known as post thrombotic syndromes. There is evidence that this may be prevented, and therefore long-term sequelae avoided, if the thrombi are dissolved quickly with thrombolytic agents. In a previous protocol we developed a method using intra-clot injections of alteplase (recombinant tissue plasminogen activator, rtPA) for the treatment of lower extremity DVT. Although the treatment was very successful with few complications, pharmacokinetic data obtained suggest that the regimen can be made safer and perhaps even more effective by using a substantially lower dose of alteplase. The current protocol is a pilot study to test this hypothesis by treating 25 patients with first-time DVT symptomatic for less than or equal to 14 days, accepted from referring physicians both within and outside the National Institutes of Health (NIH). They will be treated with less than or equal to 10 mg alteplase per day for up to four days. Depending on location and extent of the blood clot, catheters are introduced into jugular, femoral, popliteal, and/or posterior tibial vein at the ankle so as to inject alteplase (diluted with normal saline to 0.1mg/ml, throughout the entire length of the clot) once a day with each total daily dose limited to 10mg alteplase per day.The protocol is designed so that if the low-dose regimen is unsuccessful, the patient will subsequently receive the higher-dose regimen that has previously been shown to be effective. During thrombolytic therapy, catheters left in the vein to maintain venous access are also used to infuse unfractionated heparin to provide regional and therapeutic systemic anticoagulation. After completing thrombolytic therapy, the patients will be anticoagulated for approximately 6 months after treatment by conversion from intravenous infusions of unfractionated heparin during thrombolytic therapy to low molecular weight heparin (enoxaparin) and subsequent conversion to oral warfarin anticoagulation for 6 months.

Efficacy of treatments will be evaluated at 3 time points (pre- and 1 day post-thrombolytic therapy for initial outcome; at about 6 weeks for short term outcome; and at about 6 months for durability of outcome) by clinical examination (department of Rehabilitation Medicine) and medical imaging through venography and duplex ultrasound sans in department of Radiology. The protocol is also monitored for safety. Safety monitoring is focused on bleeding complications which is the primary risk of all forms of thrombolytic and anticoagulation regimens. As an adverse event, bleeding complications can be classified as either expected (for example, at vascular puncture or access sites as where treatment catheters have been inserted); or unexpected as at remote sites where no instrumentation has been conducted (for example, Intracranial or retroperitoneal bleeding).The latter form of bleeding has been reported and attributed to use of thrombolytic and anticoagulant therapies and is usually much more serious than the former. A second classification is for severity of adverse events. For this protocol a serious adverse event is an event that is life or quality of life threatening, requires additional hospitalization, or surgical intervention, or in the case of thrombolytic therapy requires blood transfusions. A minor adverse event is one that does not have any of above features and will resolve without sequelae with conservative management and without need for invasive interventions.

A secondary objective (added to this protocol through an amendment) is to study the rate of recurrent DVT during the 5 year period after treatment. Historical studies show a recurrent venothromboembolism rate of 30% in patients treated with anticoagulation alone. Thrombolytic therapy should improve preservation of venous function which may reduce recurrence rate of venothromboembolism and although the protocol cannot accrue any new patients, the protocol remains active to allow data compilation testing this hypothesis in patients already treated which will be completed by 2014, the expected date of protocol termination.

ELIGIBILITY:
INCLUSION CRITERIA

* Only adult patients (18 years old or older) are included.
* Patients must have thrombosis documented by ultrasound or venography to involve the deep veins of the pelvis and/or a lower extremity proximal to the calf veins, i.e., the popliteal vein or above.
* The thrombosis must be the patient's first DVT.
* The thrombosis must have been symptomatic for no more than 14 days.
* Patients must be able to give informed consent and be able to follow the prescribed anticoagulation regimen.
* Patients on concurrent NIH protocols will be eligible as well as patients from the community and the rest of the U.S. who are not already on NIH protocols.

EXCLUSION CRITERIA

* Pregnant patients are not eligible, although postpartum mothers over 10 days from delivery are eligible if they refrain from breast feeding their infants for 24 hours after each study with x-ray contrast material.
* Serum creatinine greater than than 2 mg/dL.
* Any current bleeding diathesis not attributable to heparin or warfarin. Fibrinogen less than 150 mg/dL. Any patient with a prothrombin time (PTT) greater than 15 s, an activated partial thromboplastin time (aPTT) greater than 35 s, or a platelet count less than 100,000/microliter must be evaluated by the Hematology Service for a coagulopathy before being included.
* Within the previous 10 days: major surgery or trauma, puncture of a noncompressible vessel, organ biopsy, or cardiopulmonary resuscitation.
* Within the previous 2 months: cerebrovascular infarction or hemorrhage, or intracranial or intraspinal surgery or trauma.
* Within the previous 6 months: major internal bleeding.
* Active intracranial disease (aneurysm, vascular malformation, neoplasm).
* Life expectancy less than 6 months.
* Patients with hemoglobin concentration less than 9g/dL will not participate in the pharmacokinetic portion of the protocol.
* Uncontrolled systolic blood pressure greater than 180 mm Hg or diastolic greater than 100 mm Hg.
* Atrial fibrillation, unless a cardiac echocardiogram excludes the presence of intracardiac thrombus.
* Known right-to-left intracardiac shunt.
* Pericarditis, infective endocarditis.
* History of heparin-induced thrombocytopenia within 6 months or the presence of persistent anti-heparin antibodies by ELISA.
* History of anaphylactic reactions to x-ray contrast media.
* Known retinopathy unless cleared by an ophthalmologist at NIH.Evidence of uncontrolled congestive heart failure or a history of diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-05; Primary Completion 2010-03 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Chang, MD, Principal Investigator — NIH Clinical Center/ Department of radiology and Imaging Sciences
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Schafer AI. Venous thrombosis as a chronic disease. N Engl J Med. 1999 Mar 25;340(12):955-6. doi: 10.1056/NEJM199903253401209. No abstract available. PMID 10089190
- [Background] Prandoni P, Lensing AW, Cogo A, Cuppini S, Villalta S, Carta M, Cattelan AM, Polistena P, Bernardi E, Prins MH. The long-term clinical course of acute deep venous thrombosis. Ann Intern Med. 1996 Jul 1;125(1):1-7. doi: 10.7326/0003-4819-125-1-199607010-00001. PMID 8644983
- [Background] Levine M, Hirsh J, Weitz J, Cruickshank M, Neemeh J, Turpie AG, Gent M. A randomized trial of a single bolus dosage regimen of recombinant tissue plasminogen activator in patients with acute pulmonary embolism. Chest. 1990 Dec;98(6):1473-9. doi: 10.1378/chest.98.6.1473. PMID 2123152
- [Background] Horne MK 3rd, Mayo DJ, Cannon RO 3rd, Chen CC, Shawker TH, Chang R. Intraclot recombinant tissue plasminogen activator in the treatment of deep venous thrombosis of the lower and upper extremities. Am J Med. 2000 Feb 15;108(3):251-5. doi: 10.1016/s0002-9343(99)00407-6. No abstract available. PMID 10723981
- [Background] Chang R, Cannon RO 3rd, Chen CC, Doppman JL, Shawker TH, Mayo DJ, Wood B, Horne MK 3rd. Daily catheter-directed single dosing of t-PA in treatment of acute deep venous thrombosis of the lower extremity. J Vasc Interv Radiol. 2001 Feb;12(2):247-52. doi: 10.1016/s1051-0443(07)61832-6. PMID 11265890
- [Result] Chang R, Horne MK 3rd, Shawker TH, Kam AW, Chen EA, Joe GO, Ching WL, Mao E, Wyrick DA Jr, Lozier JN. Low-dose, once-daily, intraclot injections of alteplase for treatment of acute deep venous thrombosis. J Vasc Interv Radiol. 2011 Aug;22(8):1107-16. doi: 10.1016/j.jvir.2011.03.023. Epub 2011 Jun 12. PMID 21664144
- [Result] Lozier JN, Cullinane AM, Nghiem K, Chang R, Horne MK 3rd. Biochemical dynamics relevant to the safety of low-dose, intraclot alteplase for deep vein thrombosis. Transl Res. 2012 Sep;160(3):217-22. doi: 10.1016/j.trsl.2012.01.025. Epub 2012 Feb 23. PMID 22683421
- [Result] Chang R, Butman JA, Lonser RR, Sherry RM, Pandalai PK, Horne MK 3rd, Lozier JN. Treatment of high-risk venous thrombosis patients using low-dose intraclot injections of recombinant tissue plasminogen activator and regional anticoagulation. J Vasc Interv Radiol. 2013 Jan;24(1):27-34.e1. doi: 10.1016/j.jvir.2012.09.017. PMID 23273695
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/B_2004-CC-0178.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in 2004 and was completed by 2009. All patients were treated at NIH Clinical Center.
Pre-assignment Details: 2 patients who were incorrectly diagnosed with Deep Vein Thrombosis (DVT) were excluded from the protocol after a preliminary ultrasound exam at NIH indicated they did not have DVT.
Groups:
- Alteplase: Dose of Alteplase will not exceed 10 mg/d/leg and is delivered in a concentration of 100ug/mL. The actual dose delivered is based upon the length of the thrombosed vein and 1 mL is injected directly into each centimeter of a thrombosed vein in a lower extremity. The treatment will be repeated up to 4 times over a 5 day period.
Period: Initial Results of Thrombolytic Therapy
Arm/Group | Alteplase
Started | 30
Completed | 28
Not Completed | 2
Not completed — died of causes unrelated to protocol | 1
Not completed — Withdrawal by Subject | 1
Period: 5 Year Recurrent Thromboembolism Rate
Arm/Group | Alteplase
Started | 28
Completed | 0 (data will not be complied until 2014)
Not Completed | 28
Not completed — will be completed 2014 | 28

BASELINE CHARACTERISTICS:
Arm/Group | Alteplase
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Restored Venous Function
Description: The outcome measures the ability of Alteplase to lyse acute and subacute deep venous thrombosis (DVT) of the lower extremities and/or pelvis and restore venous function, or blood flow, to these areas. Restored venous function is also known as patency. Patency is measured by venography and ultrasound exams.
Time Frame: 6 months
Population: The number of participants analyzed is an Intent-to-Treat (ITT) population. The initial goal was to be able to evaluate outcomes of treatment of DVT with alteplase over a 6 month period in 25 patients. 30 patients were treated but two participants did not complete the study before being assessed for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Alteplase
Number analyzed (Participants) | 30
participants | 28

2. Secondary Outcome: Number of Participants That Developed Hemorrhage
Description: The outcome measures the number of participants who developed hemorrhage after receiving up to 4 days of Alteplase treatment for DVT.
Time Frame: 5 days
Population: The number of participants analyzed is an Intent-to-Treat (ITT) population. The accrual target was to analyze outcomes(immediate, at 6 weeks, and at 6months) after treatment of DVT with alteplase in 25 patients. 30 patients were treated but two participants did not complete the study for 6 week and 6 month outcome assessments.
Measure: Number; unit: participants
Arm/Group | Alteplase
Number analyzed (Participants) | 30
participants | 0

ADVERSE EVENTS:
Time Frame: Data accumulated during 5 year study.
Arm/Group | Alteplase
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 2/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alteplase (N=30)
catheter insertion site hematoma (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Small trial of 30 patients does not have statistical power to prove clinical safety (expected to be <1 %)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes